CLINICAL TRIAL: NCT05948059
Title: A Phase I Clinical Study on Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SHR-2106 After a Single Intravenous or Subcutaneous Administration of SHR-2106 in Healthy Subjects
Brief Title: Safety and Tolerance of Increased Doses of SHR-2106 Injection in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR-2106-101
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: SHR-2106 injection or placebo single dose, iv (Experimental)
  Interventions: Drug: SHR-2106 injection or placebo
- Part 2: SHR-2106 injection or placebo single dose, sc (Experimental)
  Interventions: Drug: SHR-2106 injection or placebo

INTERVENTIONS:
Drug: SHR-2106 injection or placebo — starting dose from 50 mg
  Arms: Part 1: SHR-2106 injection or placebo single dose, iv
Drug: SHR-2106 injection or placebo — starting dose from 300 mg
  Arms: Part 2: SHR-2106 injection or placebo single dose, sc

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase I clinical study with the primary objective of evaluating the safety and tolerability of SHR-2106 in healthy subjects after a single intravenous or subcutaneous administration.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain informed consent prior to the commencement of any activities related to the trial, have a full understanding of the purpose and significance of the trial, and be willing to comply with the trial protocol;
2. Age 18 ~ 55 years old (including boundary value), male or female;
3. Male weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) = weight (kg) / height 2 (m2), BMI in the range of 19 ~ 28 kg/m2 (including boundary value);
4. Random pre-physical examination, vital signs, laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function), thyroid function, chest radiograph, 12-lead ECG results are normal or abnormal and have no clinical significance;
5. Subjects and their partners who have no fertility plan and voluntarily take highly effective contraception during the study period to the last follow-up of the trial (the last follow-up time between dose groups is shown in Table 9), 6 months (female subjects receiving SHR-2106) or 3 months (male subjects receiving SHR-2106) and voluntarily take highly effective contraception (see Annex 1 of the protocol for specific contraceptive measures), female subjects must have a negative serum pregnancy test and be non-lactating.

Exclusion Criteria:

1. The subject's medical history, symptoms and examination results at the time of screening suggest active tuberculosis or latent tuberculosis. All participants will be screened for TB status by γ interferon gamma release assay (IGRA) and chest radiograph (x-ray). Participants who underwent IGRA and x-ray examination within 1 month prior to screening may, at the discretion of the investigator, not repeat IGRA and x-ray at screening;
2. History of severe cardiovascular, liver, kidney, digestive tract, psychiatric, hematology, metabolic and other diseases (within 5 years);
3. Those who have serious infection, severe trauma or major surgery within 6 months before screening or administration; those who plan to undergo surgery during the trial;
4. Those who have chronic infection or recurrent infection within 12 months before screening and need treatment;
5. Those who donated blood or lost a total of ≥200 mL within 1 month before screening or administration, or ≥ 400 mL of blood donation or blood loss within 3 months before administration, or who received blood transfusion within 2 months;
6. Those who have a history of allergies to two or more foods and drugs; or a known history of allergy to the study drug or any component of the study drug (see Annex 2 of the protocol for injectable ingredients);
7. History of tobacco addiction within 3 months before screening, defined as: an average of more than 5 cigarettes smoked per day; or those who are unable to comply with the no-smoking requirements during the study;
8. Alcoholics within 3 months before screening (1 day intake of alcohol more than 15 g for women, more than 25 g for men [5 g of alcohol is equivalent to 150 mL of beer, 50 mL of wine or about 17 mL of low-alcohol liquor], more than 2 times a week) or positive alcohol breath test at baseline;
9. Systolic blood pressure (SBP) before screening or administration: SBP ≥ 140 mmHg or < 90 mmHg; diastolic blood pressure (DBP) :D BP≥ 90 mmHg or < 50 mmHg;
10. Glutaminase (AST) or alanine aminotransferase (ALT) at screening≥ 2 times the upper limit of normal range (ULN), or total bilirubin ≥ 1.5 times ULN
11. Those with abnormal coagulation function and clinically significant, or those who have bleeding tendency or are receiving thrombolysis or anticoagulation therapy, or those who need to receive preventive anticoagulation therapy during the test
12. Those at risk of thromboembolic events (such as history of thromboembolism, cardiovascular disease, diabetes, recurrent spontaneous miscarriage, dyslipidemia);
13. Abnormal and clinically significant 12-lead ECG results before screening or administration (e.g., male QTcF> 450 ms; QTcF for women >470 ms);
14. Those who are positive for urine drug screening during the screening period; or those with a history of substance abuse within the previous 2 years of screening;
15. Those who are positive for infectious disease screening (including hepatitis B virus surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, syphilis antibody) during the screening period;
16. Those who received live (attenuated) vaccine within 4 weeks before screening or planned to be vaccinated during the trial;
17. Those who plan to take any prescription drug, over-the-counter drug or Chinese herbal medicine that is not the test drug of the study during the screening period or 1 month before administration or within 5 half-lives of the drug (whichever is longer), or plan to take any nutritional supplement during the trial period that is not the test drug of the study (except for occasional use of acetaminophen in the recommended dose (the total amount of medication for one day does not exceed 2 g and the continuous dose does not exceed three days)) or plan to take any nutritional supplement during the trial period;
18. Those who have participated in other clinical trials or within the 5 half-lives of the investigational drug within 3 months before screening (subject to the intervention of the investigational drug or medical device, whichever is longer);
19. Have received any of the following therapies at any time: a) B-cell targeted therapy (e.g., rituximab, other anti-CD20 drugs, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], BLyS receptor fusion protein [BR3], TACI-Fc); b) Abatacept;
20. Any physical or mental illness or condition that, as determined by the study physician, may increase the risk of the trial, affect the subject's adherence to the protocol, or affect the subject's completion of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence and severity of adverse events in healthy subjects after single dose of SHR-2106 injection | About 6 months from the first medication to the evaluation

SECONDARY OUTCOMES:
Assess the concentration of SHR-2106 in plasma | About 6 months after the first dose
Evaluation of AUC0-t of SHR-2106 in plasma | About 6 months after the first dose
Evaluation of AUC0-∞ of SHR-2106 in plasma | About 6 months after the first dose
Evaluation of Tmax of SHR-2106 in plasma | About 6 months after the first dose
Evaluation of Cmax of SHR-2106 in plasma | About 6 months after the first dose
Evaluation of t1/2 of SHR-2106 in plasma | About 6 months after the first dose
To assess incidence of ADA following a single intravenous of SHR-2106 in healthy subjects | About 6 months after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- The third xiangya hospital of central south univercity, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided